CLINICAL TRIAL: NCT04034615
Title: A Phase II, Randomized, Placebo-Controlled Study of the Long-term Efficacy of Perinatal Tissue Mesenchyme Stem Cells in the Treatment for Caesarean Section Scars
Brief Title: The Long-term Effect of Perinatal Tissue Mesenchyme Stem Cells in the Treatment for Caesarean Section Scars
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The pandemic resulted in no enrollments。
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhengping Liu, MD, Director, Maternal and Child Health Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCHHFoshan-1902
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Cicatrix
Keywords: Mesenchyme Stem Cells; Cesarean Section; Scars
MeSH Terms: conditions — Cicatrix | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mesenchymal Stem Cells low-dose group (Experimental): Target dose of 3 million Mesenchymal Stem Cells
  Interventions: Biological: Mesenchyme Stem Cells low-dose group
- Mesenchymal Stem Cells high-dose group (Experimental): Target dose of 6 million Mesenchymal Stem Cells
  Interventions: Biological: Mesenchyme Stem Cells high-dose group
- Placebo (Placebo Comparator): Placebo without Mesenchyme Stem Cells
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mesenchyme Stem Cells low-dose group — Participants will receive transdermal one dose of 1*10^6 cells of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous three days and then receive transdermal placebo without of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous next three days.
  Arms: Mesenchymal Stem Cells low-dose group
Biological: Mesenchyme Stem Cells high-dose group — Participants will receive transdermal one dose of 1*10^6 cells of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous six days.
  Arms: Mesenchymal Stem Cells high-dose group
Biological: Placebo — Participants will receive transdermal placebo without of Perinatal Tissue Mesenchyme Stem Cells in the gel once a day for continuous six days.
  Arms: Placebo

SUMMARY:
The study is to investigate the long-term efficacy of perinatal tissue mesenchyme stem cells treatment on the appearance of a caesarean scar as compared to a similar untreated scar.

DETAILED DESCRIPTION:
This trial is a continuation of the investigators' previous clinical trial (NCT02772289). In the previous three-arm randomized clinical trial involving women with primiparous singleton pregnancies, the investigators found umbilical cord mesenchymal stem cells was not significantly different from placebo for the reduction of cesarean section skin scar and did not increase recognition of participants'satisfaction at the sixth month follow-up. Although there was no statistical difference, the trial study found that the total vancouver scar scale rating was lower with the dose increased.

Some studies have suggested that it usually took 18-24 months for a typical scar matures. In this trial, the investigators want to continue to investigate the efficacy of perinatal tissue mesenchyme stem cells treatment on the appearance of a caesarean scar as compared to a similar untreated scar at the three years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women receiving cesarean delivery
* Ages between 21-35 years
* Gestation ages ≥ 37 weeks and < 42 weeks
* Willing to give and sign an informed consent form and a photographic release form
* Willing to comply with study dosing and complete the entire course of the study

Exclusion Criteria:

* Any systemic uncontrolled disease
* Recent or current cancer
* History or presenting with a keloid formation
* Wounds or local disease in treatment area
* Planning any other cosmetic procedure to the study area during the study period
* Smoking

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Vancouver Scar Scale score | Three years post treatment
  The investigators measured scar at three years post treatment using Vancouver Scar Scale (VSS). The VSS included vascularity (normal, pink, red, or purple), pigmentation (normal, hypopigmented, mixed, or hyperpigmented), height (flat, < 2 mm, 2-5 mm, or > 5 mm), and pliability (normal, supple, yielding, firm, ropes, or contracture). Each variable contained ranked subscales that could be summed to obtain a total score ranging from 0 to 14, with 0 representing normal skin and a higher score representing a more marked or abnormal scar. The Chinese version of the VSS has been shown to have good intraclass correlations and Cronbach's α measures. All scars will be assessed independently by two observers on the same day when the participants are lying in a supine position with the scar exposed in bright light. If the data varies, another researcher will be required to assess the scar at the same day and the results with the highest frequency will be recorded.

SECONDARY OUTCOMES:
Erythema | Three years post treatment
  measured by reflectance
Pigmentation | Three years post treatment
  measured by reflectance
Scar Thickness and Uniformity | Three years post treatment
  A High Definition Ultrasound (US) device will be used to generate a high resolution image of the skin layers of the treated and non-treated scar in order to measure and compare changes in scar thickness and uniformity.
Subject's satisfaction | Three years post treatment
  Subject's satisfaction of the treatment using a Satisfaction Scale as follows: None; Slight; Moderate; Good; Very Good.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengping Liu, MD, Principal Investigator — Maternal and Child Health Hospital of Foshan
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China